CLINICAL TRIAL: NCT03516240
Title: The Effect of Fatigue and Biofreeze® on the Biomechanics of Running
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, Michael Holmes, Assistant Professor, Brock University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BrockURun
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants receive the topical analgesic, Biofreeze.
  Interventions: Other: Biofreeze
- Placebo (Placebo Comparator): Participants receive a placebo cream.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Biofreeze — Following a procedure that induces muscle fatigue in the lower extremity, a topical cream will be applied over the quadriceps. The cream will be either a topical analgesic (Biofreeze) or a placebo cream. Evaluation of the movement kinematics and kinetics will be evaluated for each group.
  Arms: Experimental
Other: Placebo — Following a procedure that induces muscle fatigue in the lower extremity, a topical cream will be applied over the quadriceps. The cream will be either a topical analgesic (Biofreeze) or a placebo cream. Evaluation of the movement kinematics and kinetics will be evaluated for each group. Placebo cream will be blinded to both the experimenter and study participant. It will look and smell the same and will be in the same packaging.
  Arms: Placebo

SUMMARY:
Delayed onset muscle soreness (DOMS) can be identified as the muscular pain that occurs due to intense use of skeletal muscle through exercise or other activities performed intense enough or long enough to cause minor damage(Cheung et al., 2003). DOMS usually begins to show symptoms 24 hours post-activity, becomes most intense 48-72 hours post-activity and can sometimes last up to 5-10 days in ordinary cases(Cheung et al., 2003; Dutto and Braun 2004). Typical less severe cases still can cause an individual to alter proper movement mechanics - this alteration in mechanics can lead to the further injuring of the involved or compensating skeletal muscle tissues and the associated joints and skeletal structures. DOMS-related muscular pain can lead to functional deficits and altered movement mechanics that can lead to a greater risk of further injury or sources of pain. The body does this by trying to avoid the initial source of pain by adopting some form of compensation (such as a limp when walking) which may help reduce pain at the initial source but lead to another source of pain or risk injury at another joint or limb. DOMS is a common complaint of many runners from novice to expert and due to the increased forces in running, a compensatory pattern in walking is exaggerated in running and can affect the compensating structures to an even greater extent, further increasing the risk of injury. Biofreeze®, a topical analgesic, is used to block the pain signal from the affected structures to the brain when applied to muscles experiencing delayed onset muscle soreness. Blocking the pain signal from DOMS should allow an individual to restore their natural movement mechanics.

The purpose of this study is to assess the interaction between Biofreeze® and delayed onset muscle soreness and how it affects movement mechanics and muscle function.

Hypothesis: The application of a topical analgesic (Biofreeze®) on muscles experiencing delayed onset muscle soreness (DOMS) will increase force production and return running biomechanics to pre-DOMS values.

DETAILED DESCRIPTION:
Delayed onset muscle soreness (DOMS) is a common complaint of many runners, from novice to expert. DOMS can affect the primary movers in locomotion, including but not limited to the hip flexors and extensors, knee flexors and extensors, and the ankle plantar flexors. When running with DOMS, hip, knee, and ankle mechanics can be affected in such that they may cause protective compensation in order to prevent further damage or attenuate pain in the affected musculature. One common occurrence is DOMS in the knee extensors following prolonged running. DOMS occurring in the knee extensors can greatly affect sagittal knee joint biomechanics (Dutto and Braun 2004; Paquette et al., 2017). More specifically, these changes in knee mechanics can increase knee stiffness at initial stance, resulting in an increase in vertical leg stiffness. This change in knee stiffness potentially serves as a protective compensation mechanism against lengthening of the knee extensors (Paschalis et al., 2007; Tsatalas et al., 2010). Changing running mechanics (as a result of DOMS, or fatigue) can potentially lead to an increased risk of running related injury.

One potential way to reduce or alleviate the influence of muscle soreness on running biomechanics is via topical analgesic (Ellis et al., 2005). Topical analgesics, such as Biofreeze® work by attaching to the pain receptors that transmit a signal to the brain and relay a signal back to the muscle to protect the muscle by staying in a shortened position, affecting both force production and running biomechanics (Johar et al., 2012). The blocking of this signal should allow the individual to alleviate muscular pain and return muscle function and joint mechanics to pre-DOMS levels. However, the interactive effect of muscle soreness and a topical analgesic on the biomechanics of running remains unknown. A reduction in muscular pain related to DOMS can lead to improved performance in running, or at least more comfortability in daily living when dealing with DOMS. To date, there has been little research on the interactive effect of DOMS treated with a topical analgesic on running biomechanics.

Experiment protocol

Subjects: Twenty subjects aged 17-40 years will be recruited for the study. Participants will be considered recreational runners (minimum 17 years old, running 20km per week with no recent or current injuries). Written informed consent will be obtained from all subjects.

Experimental Procedures: Before any experimental procedures, participants will be a short familiarization session and anthropometric measurements that required for motion capture analysis will be taken. Next, participants will be allowed to warm up with their regular walk/run/stretching routine. After completion, participants will be instrumented with our biomechanics equipment (see below). Next, participants will run on a treadmill. Each running session will last for 5-10 minutes and participants will run at two different speeds (2 and 3 m/s) because the effects of eccentric exercise of both knee extensors and flexors on particular tempo-spatial parameters and knee kinematics of running are speed-dependent. Following the running session at both speeds, participants will perform our DOMS protocol (see below). At 48 hours post DOMS protocol, participants will return to the lab for the exact same running protocol as described above. Next, participants will have Biofreeze® (or placebo) applied (see below) and 15 minutes following the application, participants will again perform the running protocol (see timeline below)

Day 1:

* Familiarization with protocol and lab area
* Anthropometric Measurements
* Running kinematic analysis - BASELINE (EMG and Motion Capture)
* DOMS protocol (Decline treadmill running) Day 2: (48 hours post- DOMS protocol)
* Measurement of DOMS (Pressure Pain Threshold - see appendix, Subjective Analysis)
* DOMS-induced running kinematic analysis
* Biofreeze application / Control (Placebo) application
* Intervention running kinematic analysis
* EMG and Motion Capture throughout both sessions

DOMS protocol to induce pain: The DOMS protocol will consist of participants performing a 30-minute decline treadmill running protocol. The participant will first warm up for 5 minutes at an easy walking pace on a 0% grade. Once the participant is familiar with the treadmill and is prepared, the treadmill will be set to a -10% grade (decline) and participants will work up to 85% of their predicted heart rate maximum (PHRM). Once 85% PHRM is achieved, a 30-minute timer will begin and the participant will aim to maintain that level of intensity with monitoring by a spotter that will remain by the participants side. The participant will be clipped into the safety key on the treadmill at all times when on the treadmill.

Kinematics: Three-dimensional lower body kinematics will be tracked using a 10-camera Vicon motion capture system (Vicon, Oxford, UK). Individual markers will be placed over anatomical landmarks including, medial and lateral malleoli, foot (heel, distal metatarsals), medial and lateral condyles of the knee, greater trochanters of the hip, pelvis (anterior superior iliac spines, posterior superior iliac spines), and torso (xiphoid process, suprasternal notch, T10 vertebrae, C7 vertebrae, and a medio-inferior scapular landmark for positional identification). Additionally, custom-molded rigid bodies consisting of light weight reflective markers will be secured to the dorsal surface of the foot, mid-shank laterally, mid-thigh laterally, and pelvis posteriorly (sacral-iliac region). The rigid bodies will be used to track segment movement during experimental testing. A static calibration will determine the relationship between the rigid bodies and the calibration markers over the anatomical landmarks, and subsequently joint centers and segment coordinate systems. Markers will be attached by either a velcro-nylon strap, medical tape, or double-sided tape depending on each individual location.

Electromyography (EMG): Muscle activity will be recorded using surface electromyography (SEMG) and prior to electrode placement, standard preparations, including shaving the surface and cleansing the skin with alcohol will be performed (SOP 07 - Surface EMG). The investigators will require localized shaving on the specified locations below prior to electrode placement to improve the quality of our recording sites. A single-use, disposable razor will be used and if bleeding or razor burn occurs, this will become the priority, rather than continuing the protocol. SEMG will be recorded from 8 lower extremity muscles (bilaterally). Selected muscle groups will include:

1. Knee extensors: vastus medialis, vastus lateralis, rectus femoris, vastus intermedius
2. Knee flexors: biceps femoris, semimembranosus, semitendinosus
3. Ankle plantar flexors: lateral gastrocnemius

Following electrode preparation that included shaving and scrubbing with alcohol, disposable bipolar Ag-AgCl surface electrodes (MediTrace 130, Kendall, Mansfield, MA, USA) will be placed over each muscle belly aligned with muscle fiber orientation with an interelectrode center-to-center distance of 2.5 cm. EMG will be band-pass filtered (10-1000 Hz) and differentially amplified (CMRR > 115 dB at 60 Hz; input impedance -10 GQ; Model AMT-8, Bortec Biomedical Ltd., Calgary, AB, Canada).

Following preparation, participants will perform a series of maximal voluntary contractions to normalize the EMG signals. Participants will perform isometric maximal knee flexion and extension contractions to normalize the EMG signals. All EMG data will be digitally recorded at a rate of 2048 Hz.

Pressure Pain Threshold: Pressure pain threshold will be used to assess muscle tenderness and is defined as the minimal amount of pressure that causes pain. A higher-pressure pain threshold indicates a lower amount of muscle tenderness. The pressure pain threshold will be measured for each participants' right quadricep at the beginning of each exercise session prior to any other testing. Participants will be instructed to say "yes" the instant they feel pain rather than pressure. With the participant in a relaxed standing position, the investigator will place the probe of the algometer into the midline of the right quadriceps midway between the iliac crest and the superior border of the patella. The investigator will gradually apply force at a constant rate of 50-60kPa s-1 until the participant indicates pain. Three trials, with a 30-second interval between measurement will be measured with an algometer with a 1.0cm2 stimulation area (Lafayette Instrument Company, Manual Muscle Tester, Model 01163, Lafayette, Indiana, USA.) and data will be recorded in kilograms/cm2 with a conversion to kilopascals (1kg/cm2=98.1 kPa). The average of three trials will be used for analysis.

Perceived Pain (Subjective Pain Analysis): Muscle soreness will also be measured using the BS-11 Numerical Rating Scale (NRS). The NRS will allow participants to express the amount of pain, in reference to muscle soreness they experienced. The NRS is an 11-point scale ranging 0-10, with 0 defined as "absolutely no muscle soreness", and 10 defined as "worst muscle soreness ever felt".

Rate of Perceived Exertion: A simplified scale to measure the rate of perceived exertion will be used (1-10, 1 being minimal effort and 10 being maximal effort sustainable for only a few seconds). This will be collected and averaged during every running portion of the study (Baseline, DOMS, Biofreeze/Control).

Biofreeze® (or placebo) Application: A topical cream will be applied over the quadriceps. If Biofreeze, 8ml of the topical analgesic will be applied over the muscle belly of the quadriceps. The mode of application will not involve any substantial force, pressure or rubbing, and thus any reflex activation will not be expected. This dose of Biofreeze®, is based upon the estimate that the average skin surface area over the quadriceps is approximately 1600cm2 and the recommended dosage of Biofreeze® of 1ml per 200cm. The same process will occur for the placebo cream. The researchers will be blind to application of either Biofreeze® or a placebo. Groups will be randomized into either the control or the experimental condition.

ELIGIBILITY:
Inclusion Criteria:

* Age limits
* Average 20 kilometers running per week

Exclusion Criteria:

* No recent or current injuries that would affect ability to run

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Joint angles (degrees) | 6 months
  Digitized landmarks from the trunk as well as the lower extremities will be used to create anatomical frames of reference for each modeled segment. Three-dimensional coordinates for the digitized landmarks will be continuously monitored using the fixed spatial relationship with the rigid body affixed to the segment. All kinematic data will be filtered at a rate of 6 Hz using a digital Butterworth filter. Anatomical frames of reference derived from the digitized landmarks will be used to determine joint angles in degrees throughout the selected tasks. Joint angle data will be measured for the hip, knee and ankle.
Joint velocity (degrees/second) | 6 months
  Digitized landmarks from the trunk as well as the lower extremities will be used to create anatomical frames of reference for each modeled segment. Three-dimensional coordinates for the digitized landmarks will be continuously monitored using the fixed spatial relationship with the rigid body affixed to the segment. All kinematic data will be filtered at a rate of 6 Hz using a digital Butterworth filter. Anatomical frames of reference derived from the digitized landmarks will be used to determine joint angles and velocity in degrees/second will be derived. Joint velocity data will be measured for the hip, knee and ankle.
Joint acceleration (degrees/second^2) | 6 months
  Digitized landmarks from the trunk as well as the lower extremities will be used to create anatomical frames of reference for each modeled segment. Three-dimensional coordinates for the digitized landmarks will be continuously monitored using the fixed spatial relationship with the rigid body affixed to the segment. All kinematic data will be filtered at a rate of 6 Hz using a digital Butterworth filter. Joint acceleration will be derived from joint velocity throughout the selected tasks. Joint acceleration data will be measured for the hip, knee and ankle.
Temporal measures (stride length) | 6 months
  Motion capture data will be used to determine the phase of running stride (ie. Heel strike, toe off, swing, etc.). This data will be used to determined stride length.
Temporal measures (variability) | 6 months
  Variability in stride measures throughout the repetition of the movement will be measured as a standard deviation.

SECONDARY OUTCOMES:
Muscle activity (average) | 6 months
  Average muscle activity (Surface Electromyography) will be evaluated for all muscles during all sessions. Activity will be evaluated during specific phases of a running motion. Raw signals will be full-wave rectified; digitally low-pass filtered (3Hz cut-off, 2nd order, and single pass Butterworth filtered) and normalized to the previously collected maximal voluntary contractions.
Muscle activity (maximum) | 6 months
  Maximum muscle activity (Surface Electromyography) will be evaluated for all muscles during all sessions. Activity will be evaluated during specific phases of a running motion. Raw signals will be full-wave rectified; digitally low-pass filtered (3Hz cut-off, 2nd order, and single pass Butterworth filtered) and normalized to the previously collected maximal voluntary contractions.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Holmes, PhD, Principal Investigator — Brock University
Locations (1):
- Applied Health Sciences, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dutto DJ, Braun WA. DOMS-associated changes in ankle and knee joint dynamics during running. Med Sci Sports Exerc. 2004 Apr;36(4):560-6. doi: 10.1249/01.mss.0000121957.83226.cc. PMID 15064581
- [Background] Paquette MR, Peel SA, Schilling BK, Melcher DA, Bloomer RJ. Soreness-related changes in three-dimensional running biomechanics following eccentric knee extensor exercise. Eur J Sport Sci. 2017 Jun;17(5):546-554. doi: 10.1080/17461391.2017.1290140. Epub 2017 Feb 22. PMID 28276912
- [Background] Paschalis V, Giakas G, Baltzopoulos V, Jamurtas AZ, Theoharis V, Kotzamanidis C, Koutedakis Y. The effects of muscle damage following eccentric exercise on gait biomechanics. Gait Posture. 2007 Feb;25(2):236-42. doi: 10.1016/j.gaitpost.2006.04.002. Epub 2006 May 22. PMID 16714113
- [Background] Tsatalas T, Giakas G, Spyropoulos G, Paschalis V, Nikolaidis MG, Tsaopoulos DE, Theodorou AA, Jamurtas AZ, Koutedakis Y. The effects of muscle damage on walking biomechanics are speed-dependent. Eur J Appl Physiol. 2010 Nov;110(5):977-88. doi: 10.1007/s00421-010-1589-1. Epub 2010 Jul 29. PMID 20668871
- [Background] Ellis C, Himbert A, Thompson AW, Mincer A, & Lake DA. The Effect Of Biofreeze On Delayed Onset Muscle Soreness. Journal of Orthopaedic & Sports Physical, 35(1): A34, 2005.
- [Background] Johar P, Grover V, Topp R, Behm DG. A comparison of topical menthol to ice on pain, evoked tetanic and voluntary force during delayed onset muscle soreness. Int J Sports Phys Ther. 2012 Jun;7(3):314-22. PMID 22666646
- [Background] Cheung K, Hume P, Maxwell L. Delayed onset muscle soreness : treatment strategies and performance factors. Sports Med. 2003;33(2):145-64. doi: 10.2165/00007256-200333020-00005. PMID 12617692